CLINICAL TRIAL: NCT03831295
Title: Intratumoral Injection of SD-101, an Immunostimulatory CpG Oligonucleotide, in Combination With BMS- 986178, an OX40 Agonist Antibody, in Advanced Solid Malignancies [CA012-014]
Brief Title: SD-101 and BMS-986178 in Treating Patients With Advanced or Metastatic Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald Levy (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Ronald Levy, Robert K. and Helen K. Summy Professor in the School of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-48546; NCI-2019-00251 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VAR0175 (Other: OnCore); IRB-48546 (Other: Stanford IRB)
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Extracranial Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SD-101, BMS-986178) (Experimental): SAFETY COHORT: Patients receive TLR9 agonist SD-101 IT on days 1, 8 and 15. Patients also receive anti-OX40 antibody BMS 986178 IT on days 8 and 15, and IV over 30 minutes on days 8, 29 and 58.
  EXPANSION COHORT: Patients receive TLR9 agonist SD-101 IT on days 1, 8 and 15. Patients also receive anti-OX40 antibody BMS 986178 IT on days 1, 8 and 15, and IV over 30 minutes on days 1, 29 and 58.
  Interventions: Biological: Anti-OX40 Antibody BMS 986178; Drug: TLR9 Agonist SD-101

INTERVENTIONS:
Biological: Anti-OX40 Antibody BMS 986178 — Given IT or IV
  Other Names: BMS 986178; BMS-986178
Drug: TLR9 Agonist SD-101 — Given IT
  Other Names: ISS-ODN SD-101; SD-101

SUMMARY:
This phase I trial studies the side effects of intratumoral injection of SD-101 and BMS-986178 in treating patients with solid malignancies that have spread to other places in the body. The TLR9 agonist SD-101 may stimulate the immune system in different ways and stop cancer cells from growing. BMS-986178 is a monoclonal anti-OX40 antibody that enhances the activation of T cells, immune cells that are important for fighting tumors. Giving TLR9 agonist SD-101 together with anti-OX40 antibody BMS-986178 may work better in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of intratumoral TLR9 agonist SD-101 (SD-101) in combination with intratumoral and intravenous anti-OX40 antibody BMS 986178 (BMS-986178) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

1. To evaluate the efficacy of treatment with intratumoral SD 101 in combination with intratumoral and intravenous BMS 986178 in patients with advanced solid tumors.
2. To evaluate changes in pharmacodynamic endpoints in serial tumor biopsies from I TUMOR treated and untreated sites of disease.

OUTLINE:

SAFETY COHORT: Patients receive TLR9 agonist SD-101 intratumorally (IT) on days 1, 8 and 15. Patients also receive anti-OX40 antibody BMS 986178 IT on days 8 and 15, and intravenously (IV) over 30 minutes on days 8, 29 and 58.

EXPANSION COHORT: Patients receive TLR9 agonist SD-101 IT on days 1, 8 and 15. Patients also receive anti-OX40 antibody BMS 986178 IT on days 1, 8 and 15, and IV over 30 minutes on days 1, 29 and 58.

After completion of study treatment, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Any advanced/metastatic, non-hematological, extracranial solid tumor malignancy with disease progression after at least one line of standard therapy or for which standard therapy known to prolong survival does not exist
* Patients must have at least two sites of non-osseous disease that are ≥10mm in diameter, one of which must be accessible for intratumoral injection and tumor biopsies and the other of which must be accessible for needle biopsies by interventional radiology. (Sites have to be deemed safe for repeated access upon IR review, based on anatomic location, size, shape, and accessibility). Liver lesions may not be used as the injection site even if otherwise deemed safe for access.
* Patients must have at least one additional site of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, other than the sites selected for intratumoral injection and tumor biopsies
* All patients with tumor types for which anti-PD-1 or anti PD-L1 therapy has been approved should have received such therapy prior to enrollment, with evidence of progression on at least two scans (ie, with pseudoprogression ruled out). Patients with validated driver mutations should have received and progressed on appropriate targeted therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least three months
* Total bilirubin < 1.5 x upper limit of normal (ULN) (unless patient has history of Gilbert?s disease)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN)
* Creatinine < 1.5 x ULN or measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 x ULN
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Hemoglobin >= 9 g/dL without transfusion within the past 4 weeks
* Platelets >= 100,000/mcL
* Prothrombin time (PT)/international normalized ratio (lNR) within normal limits
* Written informed consent obtained from subject
* Patients who have previously received an immune checkpoint inhibitor prior to enrollment must have any immune related toxicities resolved to =< grade 1 or baseline (prior to the checkpoint inhibitor) to be eligible. Patients who developed endocrine adverse events on checkpoint inhibitor are eligible to enter regardless of the Common Terminology Criteria for Adverse Events (CTCAE) Grade resolution as long as the patient is well controlled on endocrine replacement
* Women of childbearing potential must have a urine or serum pregnancy test within 24 hours prior to the first dose of trial treatment. If the urine test is positive or cannot be confirmed as negative, then a serum test will need to be negative
* Women of childbearing potential must practice a highly effective method of birth control during treatment and for 160 days after treatment completion. Women of childbearing potential who chose complete abstinence must agree to have a urine or serum pregnancy tests within 24h of each dose of study treatment. If the urine test is positive or cannot be confirmed as negative, then a serum test will need to be negative
* Men who are sexually active with women of childbearing potential must agree to follow instructions for methods of contraception while being treated on the study, and for 165 days after treatment completion. Men must agree to not donate sperm during this time period

Exclusion Criteria:

* History of grade 2 or higher hypersensitivity reaction to either SD-101 or BMS-986178
* Patients who require immediate treatment or cytoreduction, as deemed by their physician or the study investigators
* Treatment with other anticancer therapy (chemotherapy, small molecule, or radiation therapy) within the past 3 weeks prior to study entry or within the past 6 weeks prior to study entry for immunotherapies
* Use of investigational agent within the past 3 weeks prior to study enrollment
* Major surgery within 4 weeks of enrollment, or a wound that has not fully healed
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment
* Symptomatic central nervous system (CNS) metastases
* Known bleeding disorder that is deemed to place the patient at unacceptable risk for bleeding complications from intratumoral injection. Patients on anticoagulants and anti-platelet agents other than aspirin are excluded
* Any uncontrolled bacterial, fungal, viral, or other infection
* Active autoimmune disease requiring systemic treatment within the past 2 years, with the exception of patients well controlled on physiologic endocrine replacement
* Treatment with corticosteroids (> 10 mg per day prednisone or equivalent) or other immune suppressive drugs within 14 days prior to initiation of study drug. Steroids for topical ophthalmic, inhaled, or nasal administration are allowed. Patients requiring courses of systemic steroids for 14 consecutive days or less for an acute condition (not for a chronic autoimmune illness) may receive study drug 14 days after steroid therapy
* Prior history of cancer that is unlikely to interfere with the ability to give study treatment or affect the primary outcome or interpretation of the primary outcome of the study. For a history of malignancy treated with curative intent, enrollment should occur at least 2 years after such therapy.
* Significant cardiac disease (New York Heart Association [NYHA] class IV congestive heart failure, or unstable angina or myocardial infarction within the past 6 months)
* Human immunodeficiency virus (HIV) positive (+) patients or patients with active hepatitis B or C infection
* Patients who are pregnant or breastfeeding
* Any other medical history, including laboratory results, deemed by the investigator likely to interfere with their participation in the study, or to interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of intratumoral injections of study drugs | Up to week 96
  This outcome will be measured for any participant who has received at least one dose of any study medication. Treatment-limiting toxicities will be assessed using CTCAE v5.0. All adverse events will be recorded. Treatment-limiting toxicities are defined as;
  * Hematologic toxicities: Febrile neutropenia; Grade 3 &4 thrombocytopenia; Grade 4 anemia unexplained with exception that toxicities can clearly be determined due to disease progression and/or unrelated to SD-101 or BMS-986178.
  * Non-hematological toxicity ≥ Grade 3; Alopecia; Nausea; Grade 3 or 4 electrolyte abnormalities; Grade 3 or 4 elevation of amylase or lipase not associated with pancreatitis; Grade 3 endocrinopathy controlled by hormone replacement; Grade 3 infusion reaction that returns to Grade 1 in < 6 hours; Grade 3 skin rash not requiring systemic steroid therapy or other systemic immunosuppressive therapy.
  * Doses should be delayed if any Grade ≥ 2 toxicities are not resolved to Grade ≤ 1 or baseline by next cycle.

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years
  Tumor response assessed per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions, and assessed by physical measurement; computed tomography (CT), positron emission tomography (PET)-CT.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Progression-Free survival (PFS) | Up to 3 years
  Progression-Free Survival is defined as the time elapsed between treatment initiation (Day 1) and tumor progression or death from any cause. Progression will be defined using RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Saad A Khan, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong WX, Sagiv-Barfi I, Czerwinski DK, Sallets A, Levy R. Neoadjuvant Intratumoral Immunotherapy with TLR9 Activation and Anti-OX40 Antibody Eradicates Metastatic Cancer. Cancer Res. 2022 Apr 1;82(7):1396-1408. doi: 10.1158/0008-5472.CAN-21-1382. PMID 35135810